CLINICAL TRIAL: NCT01371266
Title: Glycemic Effects of Honey
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Grand Forks Human Nutrition Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: GFHNRC021
Record Dates: First submitted 2011-06-03; First posted 2011-06-10 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Pre-diabetes
Keywords: Glucose intolerance; Insulin resistance; Insulin; metabolic syndrome; honey; Inflammation; oxidative stress
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance; Metabolic Syndrome; Inflammation | interventions — Honey; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Honey (Active Comparator): 60.7 grams daily orally times 14 days
  Interventions: Dietary Supplement: High Fructose Corn Syrup 55 (HFCS 55); Dietary Supplement: CHO (sugar)
- CHO (Active Comparator): 50 grams daily orally times 14 days
  Interventions: Dietary Supplement: Honey; Dietary Supplement: High Fructose Corn Syrup 55 (HFCS 55)
- High Fructose Corn Syrup (Active Comparator): 65.7 grams daily orally times 14 days
  Interventions: Dietary Supplement: Honey; Dietary Supplement: CHO (sugar)

INTERVENTIONS:
Dietary Supplement: Honey — 60.7 grams orally daily times 14 days
  Arms: CHO; High Fructose Corn Syrup
Dietary Supplement: High Fructose Corn Syrup 55 (HFCS 55) — 65.7 gram daily orally times 14 days
  Arms: CHO; Honey
Dietary Supplement: CHO (sugar) — 50 grams daily orally times 14 days
  Arms: High Fructose Corn Syrup; Honey

SUMMARY:
Honey has been used as a sweetener for centuries. Recent data indicate that honey consumption may have beneficial effects upon glucose intolerance, a health issue currently affecting 57 million Americans of every age and ethnicity. In order to evaluate the glycemic effect of honey, the investigators will carry out a human trial assessing biomarkers of blood glucose responses, insulin sensitivity, oxidative stress, and inflammatory markers. Our primary objective is to determine the glycemic effects of honey in comparison to sucrose and high fructose corn syrup (HFCS). The investigators hypothesize that honey will promote improved glucose tolerance and insulin sensitivity compared to both sucrose and high fructose corn syrup in normal glycemic and glucose intolerant adults.

DETAILED DESCRIPTION:
Glucose intolerance and insulin resistance are associated with the development of the metabolic syndrome and chronic diseases, including, hyperlipidemia, hypertension, obesity, and type II diabetes. Current National Institutes of Health statistics estimate that 1 in 6 Americans have insulin resistance (www.diabetes.niddk.nih.gov/dm/pubs/statistics). Insulin resistance in humans is associated with glucose intolerance, enhanced oxidative stress, inflammation and alterations in lipid profiles. Improvements in glucose tolerance are associated with improved insulin sensitivity resulting in improved inflammatory and oxidative status. Dietary modification to reduced day-long serum insulin concentration is postulated to decrease hepatic cholesterol production through inhibition of HMG CoA reductase, the rate limiting enzyme involved in cholesterol synthesis.

Maintenance of normal blood glucose is dependent on the body's ability to modulate insulin secretion in response to the glucose load consumed. Although diet may be an important factor in glucose tolerance, the role of nutritive sweeteners has not been clearly defined. Much research has been performed on the effect of dietary sugars on chronic disease risk factors, including animal studies, and human studies ranging from epidemiologic to controlled feeding trials with most of this work focused on the monosaccharides: fructose and glucose or the disaccharide, sucrose.

Little work has been done on the comparative effects of honey and other nutritive sweeteners in relation to glucose tolerance and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women between 20-80 years of age.
2. Normal Glucose Tolerance

   * Fasting glucose between ≤105 mg/dl
   * Normal body weight or overweight (BMI 18-29.9)
3. Impaired Glucose Tolerance

   * Fasting glucose between 106-125 mg/dl
   * Overweight or obese (BMI 25 - 39.9)
4. Willingness to comply with the demands of the experimental protocol
5. Sedentary Lifestyle

Exclusion Criteria:

1. Known uncontrolled disease process
2. Diabetes mellitus
3. Use of medications that affect glucose metabolism
4. History of an eating disorder
5. Pregnancy or breast feeding
6. Inability to give consent
7. Unwillingness or inability to consume the supplemental sugars

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-06; Primary Completion 2014-12 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Area under the curve glucose, response for OGTT. Glucose-120 min OGTT-AUC | 15 weeks
  Evaluation of the effect of the treatment nutritive sweeteners on glucose tolerance.

SECONDARY OUTCOMES:
Insulin- 120 min OGTT - AUC | 15 weeks
  Evaluation of the effect of the treatment nutritive sweeteners on insulin sensitivity.
Triglycerides - 120 min OGTT - AUC | 15 weeks
  Evaluation of the effect of the treatment nutritive sweeteners on fat metabolism.
Inflammatory Markers | 15 weeks
  Effect of nutritive sweetener intake on systemic inflammation.
Oxidative Stress Markers | 15 weeks
  Effect of nutritive sweetener intake on systemic oxidative stress.
Serum Lipids | 15 weeks
  Effect of nutritive sweetener intake on lipid metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Susan K. Raatz, PhD., RD, Principal Investigator — Agriculture Research Service, United States Department of Agriculture, Grand Forks Human Nutrition Research Center
Locations (1):
- Grand Forks Human Nutrition Research Center, Grand Forks, North Dakota, United States

REFERENCES:
- [Background] Bantle JP, Raatz SK, Thomas W, Georgopoulos A. Effects of dietary fructose on plasma lipids in healthy subjects. Am J Clin Nutr. 2000 Nov;72(5):1128-34. doi: 10.1093/ajcn/72.5.1128. PMID 11063439
- [Background] Mathern JR, Raatz SK, Thomas W, Slavin JL. Effect of fenugreek fiber on satiety, blood glucose and insulin response and energy intake in obese subjects. Phytother Res. 2009 Nov;23(11):1543-8. doi: 10.1002/ptr.2795. PMID 19353539
- [Background] Raatz SK, Torkelson CJ, Redmon JB, Reck KP, Kwong CA, Swanson JE, Liu C, Thomas W, Bantle JP. Reduced glycemic index and glycemic load diets do not increase the effects of energy restriction on weight loss and insulin sensitivity in obese men and women. J Nutr. 2005 Oct;135(10):2387-91. doi: 10.1093/jn/135.10.2387. PMID 16177201
- [Background] Shah M, Adams-Huet B, Bantle JP, Henry RR, Griver KA, Raatz SK, Brinkley LJ, Reaven GM, Garg A. Effect of a high-carbohydrate versus a high--cis-monounsaturated fat diet on blood pressure in patients with type 2 diabetes. Diabetes Care. 2005 Nov;28(11):2607-12. doi: 10.2337/diacare.28.11.2607. PMID 16249527
- [Background] Andreozzi F, Laratta E, Procopio C, Hribal ML, Sciacqua A, Perticone M, Miele C, Perticone F, Sesti G. Interleukin-6 impairs the insulin signaling pathway, promoting production of nitric oxide in human umbilical vein endothelial cells. Mol Cell Biol. 2007 Mar;27(6):2372-83. doi: 10.1128/MCB.01340-06. Epub 2007 Jan 22. PMID 17242212
- [Derived] Raatz SK, Johnson LK, Picklo MJ. Consumption of Honey, Sucrose, and High-Fructose Corn Syrup Produces Similar Metabolic Effects in Glucose-Tolerant and -Intolerant Individuals. J Nutr. 2015 Oct;145(10):2265-72. doi: 10.3945/jn.115.218016. Epub 2015 Sep 2. PMID 26338891